CLINICAL TRIAL: NCT02898246
Title: Fear of Activity in Situations (FActS) - Heart Failure Study 2016
Brief Title: Fear of Activity in Situations (FActS) - Study 2016
Status: Completed | Type: Observational
Sponsor: University of Trier (Other)
Collaborators: Krankenhaus der Barmherzigen Brüder Trier (Other); Geriatric Rehabilitation Clinic St. Irminen (Other); RWTH Aachen University (Other); University Hospital, Saarland (Other)
Responsible Party: Principal Investigator, Prof. Dr. Heike Spaderna, Head of Department of Health Psychology, University of Trier
Other Study IDs: FActS Study 2016
Record Dates: First submitted 2016-09-02; First posted 2016-09-13 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Chronic Heart Failure; Fear of Movement (Fear of Physical Activity)
Keywords: heart failure; fear of physical activity; motor activity
MeSH Terms: conditions — Kinesiophobia; Heart Failure; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with chronic heart failure: Fear of physical activity (exposure) will be assessed in adult outpatients with diagnosed, chronic heart failure (with reduced ejection fraction or with preserved ejection fraction).
  Hospitals provide medical data to assess patients' disease severity. Additional measures assessed via questionnaire include demographic characteristics, State and Trait depression and anxiety, heart failure related symptom distress, and coping dispositions relevant for coping with physical threat.
  Fear of physical activity (FActS-HF 15) is reassessed after 4 weeks to evaluate the instrument's retest reliability.
  After questionnaire completion, a subsample of participants will wear the MOVE III accelerometer for one week to objectively assess everyday physical activity and fill in an activity diary.

SUMMARY:
The aim of the study is to evaluate the psychometric properties of the newly developed Fear of Activity in Situations - Heart Failure (FActS-HF 15) scale. The FActS-HF 15 is a questionnaire assessing fear of physical activity (fear of movement) in patients with chronic heart failure. FActS-HF 15 assesses cognitions and emotions that can occur during physical activity, independent of avoidance behavior. Firstly, the study aims at evaluating the instrument's reliability and validity and to investigate associations of fear of physical activity with demographic, medical, and psychosocial patient characteristics. Secondly, the study aims at assessing everyday physical activity using accelerometric measures to test the hypothesis that fear of physical activity in patients with heart failure is related with lower actual physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of heart failure stage B or C (Hunt et al., 2005), or: New York Heart Failure classification II to IIIb:

  1. Systolic dysfunction: left ventricular ejection fraction < 45% in the last 6 month
  2. Diastolic dysfunction: left ventricular ejection fraction >= 45% in the last 6 month

Exclusion Criteria:

* complex ventricular arrhythmias
* acute myocarditis
* symptomatic cardiac valve stenosis
* instable angina pectoris
* other severe diseases, that impair physical activity (e.g., advanced stages of cancer)
* insufficient language skills in German to answer the questionnaires
* insufficient cognitive skills to answer the questionnaires

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients with diagnosed chronic heart failure of all underlying diagnoses. Patients have to be outpatients at time of study participation. They will be recruted in primary care clinics, and heart failure outpatient clinics in Germany.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2016-11; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
FActS-HF 15 total score and subscores | 2016-2019
  The psychometric properties of FActS-HF 15 are assessed in terms of item analysis, reliability (internal consistency, test-retest reliability), convergent and discriminant validity (correlations with other questionnaires) as well as confirmatory factor analysis (assessing the dimensionality). Associations with demographic, medical, and psychosocial variables will be evaluated.

SECONDARY OUTCOMES:
Average daily energy expenditure due to physical activity (kcal/d) | 6 day assessment, after questionnaire completion
  Objectively assessed via accelerometry
Average intensity of physical activity (MET) | 6 day assessment, after questionnaire completion
  Objectively assessed via accelerometry
Average relative frequency of activity classes | 6 day assessment, after questionnaire completion
  Relative frequency of activity classes stair climbing, lying down, walking

CONTACTS AND LOCATIONS:
Overall Officials: Heike Spaderna, PhD, Principal Investigator — Trier University
Locations (6):
- Germany (6):
  - Universitätsklinikum Aachen, Aachen
  - Universitätsklinikum des Saarlands, Homburg
  - Mutterhaus der Borromäerinnen, Trier
  - Geriatrische Rehabilitationsklinik St. Irminen, Trier
  - Krankenhaus der Barmherzigen Brüder Trier, Trier
  - Rhein-Maas-Klinikum, Würselen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luke T, Brandenburg VM, Partetzke TM, Voss F, Spaderna H. Accelerometer-Measured Daily Physical Activity in Adults With Chronic Heart Failure and Associations With Fear of Physical Activity and Coping Dispositions. J Cardiovasc Nurs. 2025 Jul 28. doi: 10.1097/JCN.0000000000001242. Online ahead of print. PMID 40719556
- [Derived] Spaderna H, Brandenburg VM, Lauterbach M, Partetzke TM, Schwab SU, Voss F, Kindermann I. Associations of fear of physical activity, coping style and self-reported exercise behavior in patients with chronic heart failure. PLoS One. 2024 Sep 5;19(9):e0309952. doi: 10.1371/journal.pone.0309952. eCollection 2024. PMID 39236063